CLINICAL TRIAL: NCT00223626
Title: Lab Trials to Develop Medication for Cocaine Dependence
Brief Title: Topiramate to Reduce Cocaine Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bankole Johnson (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Bankole Johnson, Chair of Psychiatry and Neurobehavioral Sciences, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 12350; R01DA012191 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Cocaine-Related Disorders
Keywords: Cocaine Addiction; Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental)
  Interventions: Drug: Topiramate
- Placebo (Placebo Comparator)
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — the maximum topiramate test dose is 200 mg/d.
  Other Names: Topamax

SUMMARY:
Cocaine addiction is a serious health problem with no available medical treatment for preventing relapse. Topiramate, a medication which lowers dopamine levels, may have the ability to diminish cocaine cravings in addicts. The purpose of this study is to determine the effectiveness of topiramate in reducing cocaine's rewarding effects in individuals addicted to cocaine.

DETAILED DESCRIPTION:
GABA is an inhibitory neurotransmitter that is found primarily in the brain. High GABA levels result in low levels of dopamine, another neurotransmitter that is the brain's "feel good" chemical and which plays a primary role in cocaine drug addiction. Cravings for cocaine can be reduced by lowering dopamine levels. This makes topiramate, a GABA-altering medication, a potential treatment for cocaine addiction. This study will evaluate the subjective, behavioral, and physiological effects of topiramate in individuals addicted to cocaine.

Potential participants will initially attend a 4- to 6-hour screening session. This will include review of medical and drug histories, standardized psychological questionnaires, a physical exam, and blood collection. Eligible participants will then be admitted to the inpatient clinic. During the first day of experiment, participants will receive instructions and information about the study procedures. They will also undergo a physical exam, an electrocardiogram, standardized psychological questionnaires, and blood and urine collection. A single test dose of cocaine will be administered intravenously to all participants to ensure safety with continuation in the study. Vital signs will be monitored hourly throughout the day.

The experiment will last 25 days and will enroll 24 individuals addicted to cocaine. In this three-part experiment, participants will be admitted to the inpatient clinic for an 8-day study session. Following this session, they will be discharged from the clinic for a 1-week washout phase. Participants will then return to the inpatient clinic for another 8-day study session. The two study sessions will be identical. During both sessions, participants will first receive topiramate or placebo for 4 consecutive days. While continuing to receive topiramate or placebo, participants will then also receive intravenous cocaine or placebo for 3 consecutive days.Participants will be monitored by the study physician. Electrocardiograms will be used to monitor heart activity, and blood will be drawn frequently to monitor levels of cocaine and topiramate. Participants will complete standardized questionnaires several times each day to assess mood changes and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV-TRTM diagnostic criteria for cocaine dependence
* Subjects must be non-treatment seeking, cocaine-dependent or cocaine-abusing individuals who report taking cocaine at least once a month
* In generally good health as confirmed by medical history, physical examination, electrocardiogram, laboratory screening tests, and vital signs
* Must be able to take oral medication, adhere to the medication regimens, and be willing to return to the clinic for regular study visits
* Must be able to read and understand all instructions, rating scales, and questionnaires in English
* Must be willing to stay overnight at the University Clinical Psychopharmacology Laboratory (UCPL)
* Must comply with the alcohol, tobacco, and drug-free environment regulations at the UCPL
* If female, must be postmenopausal for at least 1 year, surgically sterile, or willing to use contraception throughout the study

Exclusion Criteria:

* History of mental illness, other than cocaine or nicotine dependence
* History of mental retardation or neuropsychological functioning greater than 1.5 standard deviation below expected rang.
* Clinically significant abnormalities found on the electrocardiogram
* History of hypertension (blood pressure greater than 140/90 mm Hg) or systolic hypotension (blood pressure less than 90/75 mm Hg)
* Resting pulse rate of greater than 90 beats per minute
* Cerebrovascular accident or transient ischemic attack
* Ischemic heart disease or heart attack
* Symptomatic coronary artery disease or peripheral vascular disease
* Cancer or history of cancer within the 5 years of study entry (other than basal cell carcinoma)
* Kidney disease and/or impaired kidney function, as defined by an estimated creatinine clearance of 60 mL per minute
* Gastrointestinal system disease, including active liver disease or current active hepatitis; subjects with AST and/or ALT levels greater than four times the upper limit of the normal range and/or an increased total serum bilirubin level greater than two times the upper limit of normal at screening
* Endocrinological disorders, including thyroid disorders
* Glaucoma
* Gross neurological disorders, including seizure disorders and progressive or degenerative neurological disorders (e.g., multiple sclerosis)
* History of nephrolithiasis
* Clinically significant laboratory screening test results on hematology, chemistry, or urine analysis; up to four times above the normal range of the following will be allowed unless there is evidence of hepatocellular disease or failure: liver enzymes (SGOT), serum glutamic pyruvic transaminase (SGPT), gamma-glutamyltransferase (GGT), blood urea nitrogen (BUN), lactate dehydrogenase (LDH)
* Any disease or condition that compromises the function of body systems that may result in altered absorption, excess accumulation, or impaired metabolism or excretion of topiramate
* Current use of psychoactive drugs, including sympathomimetics, caffeinated drinks in excess of 500 mg per day, and tobacco consumption of greater than 0.75 grams per day (approximately 25 cigarettes per day); non-pathological levels of alcohol consumption is permitted
* Suicide attempt or suicidal thoughts within 30 days of study entry
* Evidence of behavioral toxicity, including seizures, severe agitation, or psychosis
* Be taking a medication that could interact adversely with topiramate, unless the medication is discontinued.
* History of any severe or life-threatening medication interactions
* Currently taking any prescribed medications for heart or cerebrovascular disease
* Currently taking any medication with potential interactions with cocaine or topiramate, including glutamate antagonists (e.g., acamprosate), serotonin re-uptake inhibitors (e.g., fluoxetine), serotonin antagonists (e.g., ritanserin or buspirone), other antidepressants (e.g., tricyclic antidepressants or monoamine oxidase inhibitors), dopamine antagonists (e.g., haloperidol), calcium channel antagonists (e.g., isradipine), compounds with actions similar to disulfiram (Antabuse), or any carbonic anhydrase medication or medication containing triamterene
* Previously treated with topiramate for any reason and discontinued treatment due to an adverse event or a hypersensitivity reaction to topiramate
* Participation deemed unsafe because of precautions, warnings, or contraindications outlined in the topiramate investigator brochure and/or package insert, as determined by study investigator
* Expected to stay in a restricted environment or awaiting imprisonment
* Currently living in the same household as another study participant
* Received an investigational drug or device or participated in a clinical trial in the 30 days prior to study entry
* Employee of the investigator or study center
* Pregnant or breastfeeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cocaine-induced mood changes | measured throughout cocaine and topiramate testing sessions
Effects of topiramate on cognitive function | measured throughout cocaine and topiramate testing sessions
Drug safety | measured throughout cocaine and topiramate testing sessions
Cardiovascular response to cocaine (measured throughout cocaine and topiramate testing sessions) | measured throughout cocaine and topiramate testing sessions

SECONDARY OUTCOMES:
Physiological response (measured throughout cocaine and topiramate testing sessions) | measured throughout cocaine and topiramate testing sessions

CONTACTS AND LOCATIONS:
Overall Officials: Bankole A. Johnson, DSc,MD.PhD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia CARE Center for Addiction Research & Education, Charlottesville, Virginia
  - UVA CARE Richmond, Richmond, Virginia